CLINICAL TRIAL: NCT01255670
Title: Penicillin and Metronidazole in Treatment of Peritonsillar Abscess - Prospective, Double-blind, Randomized, Placebo-controlled Study
Brief Title: Penicillin and Metronidazole in Treatment of Peritonsillar Abscess
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Karin Blomgren, Senior Medical Officer in Charge of Research, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 224/13/03/02/2009
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Peritonsillar Abscess
Keywords: Peritonsillar Abscess; Quinsy; Penicillin; Metronidazole; Recurrence
MeSH Terms: conditions — Peritonsillar Abscess; Recurrence | interventions — Penicillins; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- penicillin and metronidazole (Active Comparator): After incision and drainage 100 randomized patients receive penicillin and metronidazole as treatment of peritonsillar abscess
  Interventions: Drug: penicillin and metronidazole in peritonsillar abscess
- penicillin and placebo (Placebo Comparator): After incision and drainage 100 randomized patients receive penicillin and placebo as treatment of peritonsillar abscess
  Interventions: Drug: penicillin and metronidazole in peritonsillar abscess

INTERVENTIONS:
Drug: penicillin and metronidazole in peritonsillar abscess — Peroral Penicillin: 1000 000 IU 3 times a day for 10 days Peroral metronidazole: 500 mg 3 times a day for 7 days
  Other Names: Medicillin; Flagyl; Tricozol

SUMMARY:
Treatment of peritonsillar abscess varies. To study whether broad spectrum antibiotics are required in addition to abscess drainage, a prospective, double blind, placebo-controlled, randomized study on 200 adult patients with peritonsillar abscess is performed. 100 patients are given penicillin and metronidazole and 100 patients get penicillin and placebo. Recovery and recurrence are analyzed.

ELIGIBILITY:
Inclusion Criteria:

* referring doctor suspects peritonsillar abscess
* patient is voluntary
* patient has daily access to his/her e-mail
* patient speaks and understands Finnish of Swedish
* female patients have adequate birth-control method
* patient has peritonsillar abscess

Exclusion Criteria:

* allergy to penicillin
* allergy to metronidazole
* use of metronidazole in preceding one month
* pregnancy
* breast-feeding
* renal insufficiency
* liver insufficiency
* alcoholism (drunk at least once a week)
* participant in another clinical trial at the moment
* treatment of peritonsillar abscess requires in-patient care
* tonsillectomy during the next 30 days
* army recruit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin V Blomgren, MD, PhD, Principal Investigator — consultant
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wiksten JE, Pitkaranta A, Blomgren K. Metronidazole in conjunction with penicillin neither prevents recurrence nor enhances recovery from peritonsillar abscess when compared with penicillin alone: a prospective, double-blind, randomized, placebo-controlled trial. J Antimicrob Chemother. 2016 Jun;71(6):1681-7. doi: 10.1093/jac/dkw038. Epub 2016 Mar 10. PMID 26968881

RESULTS

PARTICIPANT FLOW:
Groups:
- Penicillin and Metronidazole: After incision and drainage 100 randomized patients receive penicillin and metronidazole as treatment of peritonsillar abscess.
  Penicillin and metronidazole in peritonsillar abscess: Peroral Penicillin: 1000 000 IU 3 times a day for 10 days; Peroral metronidazole: 500 mg 3 times a day for 7 days.
- Penicillin and Placebo: After incision and drainage 100 randomized patients receive penicillin and placebo as treatment of peritonsillar abscess.
  Penicillin and metronidazole in peritonsillar abscess: Peroral Penicillin: 1000 000 IU 3 times a day for 10 days; Peroral metronidazole: 500 mg 3 times a day for 7 days.
Period: Overall Study
Arm/Group | Penicillin and Metronidazole | Penicillin and Placebo
Started | 100 | 100
Completed | 74 | 80
Not Completed | 26 | 20
Not completed — Adverse Event | 10 | 10
Not completed — Lost to Follow-up | 16 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Penicillin and Metronidazole | Penicillin and Placebo | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 100 | 100 | 200
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 44 | 91
  Male | 53 | 56 | 109
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Finland | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Recurrence of Peritonsillar Abscess
Description: Number of participants with recurrence of peritonsillar abscess having metronidazole in addition to penicillin or penicillin and placebo.
Time Frame: 56 days
Measure: Count of Participants; unit: Participants
Arm/Group | Penicillin and Metronidazole | Penicillin and Placebo
Number analyzed (Participants) | 100 | 100
Participants | 10 | 10
Statistical Analysis 1: Comparison: Penicillin and Metronidazole vs Penicillin and Placebo; Test type: Other — Mann-Whitney U-test and Fisher's exact test; p = 0.05, Fisher Exact

2. Secondary Outcome: Number of Participants Recovering From Peritonsillar Abscess
Description: Number of participants recovering from peritonsillar abscess having metronidazole in addition to penicillin or penicillin and placebo.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Penicillin and Metronidazole | Penicillin and Placebo
Number analyzed (Participants) | 84 | 90
Participants | 74 | 80
Statistical Analysis 1: Comparison: Penicillin and Metronidazole vs Penicillin and Placebo; Mann-Whitney U-test and Fisher's exact test; Test type: Other; p = 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Penicillin and Metronidazole | Penicillin and Placebo
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 61/100 | 51/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Penicillin and Metronidazole (N=100) | Penicillin and Placebo (N=100)
Nausea (Gastrointestinal disorders) | 10 | 8
Diarrhea (Metabolism and nutrition disorders) | 16 | 10
Dizziness (Nervous system disorders) | 12 | 16
Headache (Nervous system disorders) | 15 | 12
Rash (Skin and subcutaneous tissue disorders) | 8 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes